CLINICAL TRIAL: NCT02770495
Title: Dynamics of Regulatory and Effector T Lymphocyte Subsets in Patients With Crohn's Disease During Postoperative Recurrence : Implications for Identifying Patients at High Risk of Relapse.
Brief Title: Postoperative REcurrence and DynamICs of T Cell Subsets in Crohn's Disease
Acronym: PREDICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-616
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Postoperative endoscopic recurrence (Experimental): Patients with a diagnosis of Crohn's disease who undergo an ileo-colonic curative resection
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
It is assumed that gut inflammation and lesions characterizing flares of Crohn's disease (CD) result from an aberrant T-cell mediated immune responses characterized by a complex balance between peripheral and lamina propria regulatory and effector T cell subsets. Because most of CD patients who undergo a surgery experienced a postoperative endoscopic recurrence of the disease (70 % at one year) leading to a clinical recurrence (10 % per year), the "model" of postoperative recurrence in CD represents a privileged situation that mimicks what happens in the gut of CD patients in clinical remission before the occurrence of further flares. It is likely that the same factors which underlie the immunopathogenesis of CD at its early stages also contribute to disease recurrence in the postoperative setting. Indeed, the postoperative state is performed for intent of disease remission and this situation represents probably an ideal setting to investigate the dynamics of most of T cell subsets in the peripheral and mucosal compartments because one may argue that removal of the diseased segment of bowel resets the disease to its earliest phases, providing an interesting window to better understand which T cell subsets predispose to disease recurrence.

That is the reason why this model will be used in the present project i) to understand better the immunopathogenesis of CD relapse; ii) to identify novel and promising immune cell-associated biomarkers capable to predict relapse of the disease and finally iii) to identify potential specific therapeutic target associated with T cell subsets involved in the initiation of disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Men or non-pregnant women
* Patients with a diagnosis of Crohn's disease who undergo an ileo-colonic curative resection
* No change of the postoperative treatment before assessing an endoscopic recurrence during the one-year post surgery follow-up period
* Informed consent given

Exclusion Criteria:

* Pregnancy
* History of disease, including mental/emotional disorder, that might interfere with their participation in the study
* Inability to comply with the protocol requirements
* Inability to fill in the diary cards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Postoperative endoscopic recurrence, assessed by a Rutgeerts 's score > i1, over the one-year post-surgery follow-up | at one year
  Rutgeerts 's score > i1

SECONDARY OUTCOMES:
proportion of T cell subsets in the arm of patients who will experience a recurrence and those who will not. | at 3 months before relapse
number of T cell subsets in the arm of patients who will experience a recurrence and those who will not. | at 3 months before relapse

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane NANCEY, MD, Principal Investigator — Service d'Hépato-Gastroentérologie Centre hospitalier Lyon Sud Hospices Civils de Lyon
Locations (1):
- Service d'Hépato-Gastroentérologie Centre hospitalier Lyon Sud Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Result] Boschetti G, Nancey S, Moussata D, Cotte E, Francois Y, Flourie B, Kaiserlian D. Enrichment of Circulating and Mucosal Cytotoxic CD8+ T Cells Is Associated with Postoperative Endoscopic Recurrence in Patients with Crohn's Disease. J Crohns Colitis. 2016 Mar;10(3):338-45. doi: 10.1093/ecco-jcc/jjv211. Epub 2015 Nov 19. PMID 26589954